CLINICAL TRIAL: NCT04935229
Title: A Phase 1/1b, Open-Label Study of the Pressure-Enabled Hepatic Artery Infusion of SD-101, a TLR9 Agonist, Alone or in Combination With Intravenous Checkpoint Blockade in Adults With Metastatic Uveal Melanoma
Brief Title: Intrahepatic Delivery of SD-101 by Pressure-Enabled Regional Immuno-oncology (PERIO), With Checkpoint Blockade in Adults With Metastatic Uveal Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision was made to terminate the study after the completion of Phase 1 enrollment and not proceed with Phase 2. Trial termination was not due to patient safety or data concerns.
Sponsor: TriSalus Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS-PERIO-01
Record Dates: First submitted 2021-06-02; First posted 2021-06-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Uveal Melanoma in the Liver
Keywords: Uveal Melanoma; Liver Metastases; TLR9; SD-101
MeSH Terms: conditions — Uveal Melanoma | interventions — Nivolumab; Ipilimumab; relatlimab; Opdualag

STUDY DESIGN:
Intervention Model Description: Sentinel Cohort: Two doses of SD-101 (0.5mg and 2mg) administered 2 weeks apart via PEDD/HAI using the TriNav device.
  Cohorts A, B, C, and Phase 1b: Three weekly doses of SD-101 (given over two 52-day cycles) in dose-escalation fashion (2mg, 4mg, 8mg-optional) via PEDD/HAI using the TriNav device.
  Cohort D (optional): Two weekly doses of SD-101 (given over two 52-day cycles) via PEDD/HAI using the TriNav device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SD-101 (Experimental): 3 weekly doses of SD-101 given via hepatic artery infusion over 2 cycles
  Interventions: Drug: SD-101; Biological: Nivolumab; Biological: Ipilimumab; Biological: Nivolumab and Relatlimab

INTERVENTIONS:
Drug: SD-101 — SD-101 doses will be delivered via hepatic artery infusion using pressure enabled drug delivery using the TriNav device
Biological: Nivolumab — During Cohort B, nivolumab will be administered together with SD-101 and during Cohort C, it will be administered with ipilimumab and SD-101
  Other Names: Opdivo
Biological: Ipilimumab — During Cohort C, ipilimumab will be administered together with nivolumab and SD-101
  Other Names: Yervoy
Biological: Nivolumab and Relatlimab — During optional Cohort C1, nivolumab and relatlimab will be administered with SD-101
  Other Names: Opdualag

SUMMARY:
This study is an open-label, phase 1/1b study of the pressure-enabled hepatic artery infusion of SD-101, a TLR 9 agonist, alone or in combination with intravenous checkpoint blockade in adults with metastatic uveal melanoma.

DETAILED DESCRIPTION:
In the Sentinel Cohort, patients will receive 2 SD-101 infusions (2 weeks apart) with assessments for toxicity prior to escalating from the first dose level (0.5 mg) to the second dose level (2 mg). In the absence of dose-limiting toxicities (DLTs), each patient will be eligible to transition into Cohort A.

In Cohorts A-C and Phase 1b, patients will receive 2 cycles of SD-101. Each cycle consists of 3 consecutive weekly infusions. Escalating doses of SD-101 will be administered alone (Cohort A), together with nivolumab (Cohort B), together with combined ipilimumab and nivolumab (Cohort C), or together with nivolumab and relatlimab (Cohort C1 - optional). Cohorts B and C will begin dosing at the minimum anticipated biological effect level (MABEL(2mg SD-101)).

An optional Cohort D may be opened to explore the combination of one or more of the following three CPI regimens with a modified SD-101 dosing schedule with only 2 weekly SD-101 infusions per cycle for 2 cycles:

1. Single-agent nivolumab IV at 480mg every 4 weeks;
2. IV ipilimumab 3mg/kg and IV nivolumab 1mg/kg every 3 weeks for 4 doses each followed thereafter by nivolumab 480mg IV every 4 weeks;
3. Nivolumab 480mg and relatlimab 160mg IV every 4 weeks.

Following determination of the recommended MTD or optimal dose of SD-101 for PEDD/HAI and which checkpoint inhibitor (CPI) regimen(s) are tolerated, the study will progress to Phase 1b. Patients in Phase 1b will receive the SD-101 dose selected from Phase 1 together with systemic single- or double-agent checkpoint blockade. The choice of single- or double-agent CPI therapy together with SD-101 for Phase 1b will consider safety data in addition to response rates from Cohorts B and C in Phase 1.

Patients enrolled into the main study are eligible to enroll into an optional imaging sub-study investigating the use of 89Zr-Df-crefmirlimab, a biologic PET radioligand for detecting CD8+ T cell lymphocytes. 89Zr-Df-crefmirlimab will be administered by IV at screening and again prior to C2D1 procedures. A PET scan is conducted within 72 hours following the tracer infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years of age at screening
2. Able to understand the study and provide written informed consent prior to any study procedures
3. Has histologically or cytologically confirmed metastatic UM with liver-only or liver dominant disease. Liver-dominant disease will be defined as intrahepatic metastases representing the largest fraction of disease relative to other organs.
4. Has not received prior cytotoxic chemotherapy, targeted therapy, or external radiation therapy within 14 days prior to screening
5. Has not received therapy with prior immunological checkpoint blockade within 21 days before the first dose of study intervention and has no ongoing immune-mediated AEs Grade 2 or higher
6. Has not ever received prior embolic HAI therapy with permanent embolic material Note: Previous embolic HAI therapy with permanent embolic material will not be exclusionary if following this therapy, the target vessels are not occluded and the liver segments containing target tumors are perfused based on the patient's screening CT/MRI.
7. Prior surgical resection or radiofrequency ablation of oligometastatic liver disease is allowed on both the Phase 1 and Phase 1b portions of this study. Liver lesions that received ablative therapies should not be considered target lesions unless they have clearly progressed since the therapy.
8. Has no prior history of or other concurrent malignancy unless the malignancy is clinically insignificant, no ongoing treatment is required, and the patient is clinically stable
9. Has measurable disease in the liver according to RECIST v.1.1 criteria
10. Has an ECOG PS of 0-1 at screening
11. Has a life expectancy of >3 months at screening as estimated by the investigator
12. Has a QTc interval ≤480 msec
13. All associated clinically significant (in the judgment of the investigator) drug-related toxicity from previous cancer therapy must be resolved (to Grade ≤1 or the patient's pretreatment level) prior to study treatment administration (Grade 2 alopecia and endocrinopathies controlled on replacement therapy are allowed)
14. Has adequate organ function at screening as evidenced by:

    * Platelet count >100,000/μL
    * Hemoglobin ≥8.0 g/dL
    * White blood cell count (WBC) >2,000/μL
    * Serum creatinine ≤2.0 mg/dL unless the measured creatinine clearance is ≥30 mL/min calculated by Cockcroft-Gault formula.
    * Total and direct bilirubin ≤2.0 × the upper limit of normal (ULN) and alkaline phosphatase ≤5 × ULN. For patients with documented Gilbert's disease, total bilirubin up to 3.0 mg/dL is allowed.
    * ALT and AST ≤5 × ULN
    * Prothrombin time/International Normalized Ratio (INR) or activated partial thromboplastin time (aPTT) test results at screening ≤1.5 × ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose for at least 4 weeks prior to the first dose of study intervention) Note: Laboratory tests with exclusionary results judged by the investigator as not compatible with the patient's clinical status may be repeated once for eligibility purposes.
15. Females of childbearing potential must be nonpregnant and nonlactating, or post-menopausal, and have a negative serum human chorionic gonadotropin (hCG) pregnancy test result at screening and a negative urine or serum pregnancy test prior to the first dose of study intervention.

    * Females of childbearing potential must agree to abstain from sexual activity with nonsterilized male partners, or if sexually active with a nonsterilized male partner must agree to use highly effective methods of contraception from screening, throughout the study and agree to continue using such precautions for 100 days after the final dose of study intervention.
    * Nonsterilized males who are sexually active with a female of childbearing potential must agree to use effective methods of contraception and avoid sperm donation from Day 1, throughout the study, and for 30 days after the final dose of study intervention.

Exclusion Criteria:

1. Has received chemotherapy or an investigational agent within 14 days (or 5 half-lives, whichever is shorter) before screening
2. Has active, untreated brain metastasis
3. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
4. Has portal vein thrombosis, or severe portal hypertension as defined by a history of variceal hemorrhage or active ascites accumulation
5. Has more than 2/3 parenchymal replacement by tumor of both liver lobes
6. Phase 1 and Phase 1b:

   1. Has Child-Pugh Class B or C cirrhosis, or
   2. Has experienced a Grade 3 or higher immune-related AE from prior CPI therapy that has not recovered to Grade 1 for a minimum of 14 days prior to administration of SD-101 or CPI, or
   3. Is unable to be temporarily removed from chronic anticoagulation therapy, or
   4. Has a history of bleeding disorders
7. Has active coronavirus disease 2019 (COVID-19), other severe infection, including a liver infection, within 2 weeks before the first dose of study drug, or uncontrolled human immunodeficiency virus (HIV) infection at screening
8. Has had bacterial pneumonia within 8 weeks of first dose of study drug
9. Has active, known, or suspected autoimmune disease or immune-mediated disease. Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment or conditions not expected to recur in the absences of an external trigger are not exclusionary.
10. Is receiving systemic steroid therapy >10 mg of prednisone daily or equivalent or any other immunosuppressive medication at any dose level. Local steroid therapies (e.g., otic, ophthalmic, intra-articular or inhaled medications) are acceptable.
11. Has significant concurrent or intercurrent illness, psychiatric disorder, or alcohol or chemical dependence that would, in the opinion of the Investigator and/or Medical Monitor, compromise their safety or compliance or interfere with interpretation of the study
12. Lactating women are excluded from study participation
13. Has previously received SD-101
14. Medical history of significant hypersensitivity, severe and unresolved immune-mediated reactions, severe infusion-related reactions, or allergic reaction to TLR9 agonists or CPI agents in the judgment of the investigator
15. Patients who were enrolled in the Phase 1 portion of the study will not be eligible for enrollment in Phase 1b

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Phase 1: To Determine the Safety of SD-101 Alone, in Combination with Nivolumab, and in Combination with Both Nivolumab and Ipilimumab | 12 months
  As a measure of safety, adverse events will be graded according to CTCAE v5.0.
Phase 1: To Determine the Maximum Tolerable Dose (MTD) or Optimal Dose of SD-101 alone, in Combination with Nivolumab, and in Combination with Both Nivolumab and Ipilimumab | 12 months
  A standard 3+3 dose-escalation design will be employed to determine the MTD or optimal dose.
Phase 1b: To Assess Overall Response Rate (ORR) | 12 months
  As a measure of activity, ORR will be assessed. ORR will be assessed using Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
Phase 1b: To Assess Overall Survival (OS) | 12 months
  As a measure of activity, OS will be assessed. The events for the assessment of 12-month OS are death events.

SECONDARY OUTCOMES:
Phase 1: Determination of Single vs. Dual-agent CPI in Phase 1b using CTCAE v5.0 | 6 months
  The choice of single- or dual-agent CPI therapy together with SD-101 for Phase 1b will consider AEs/SAEs per CTCAE v5.0.
Phase 1: Determination of Single vs. Dual-agent CPI in Phase 1b using RECIST v1.1 | 6 months
  The choice of single- or dual-agent CPI therapy together with SD-101 for Phase 1b will consider response rates per RECIST v1.1 from Cohorts B and C in Phase 1.
Phase 1b: To Assess Treatment-Emergent Adverse Events of the Chosen MTD or Optimal Dose of SD-101 in Combination with CPI | 6 months
  As a measure of safety, adverse events will be graded according to CTCAE v5.0.
Phase 1b: Assess Preliminary Efficacy in Terms of iRECIST for Immune Based Therapeutics | 12 months
  As a measure of activity, iRECIST will be utilized to determine ORR.
Phase 1b: Assess Preliminary Efficacy in Terms of modified RECIST (mRECIST) for Immune Based Therapeutics | 12 months
  As a measure of activity, mRECIST will be utilized to determine ORR.
Phase 1b: Assess Preliminary Efficacy in Terms of RECIST v1.1 for Immune Based Therapeutics | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine hepatic-specific response rate (HRR).
Phase 1b: Assess Preliminary Efficacy in Terms of RECIST v1.1 for Immune Based Therapeutics | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine duration of response (DOR).
Phase 1b: Assess Preliminary Efficacy in Terms of RECIST v1.1 for Immune Based Therapeutics | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine overall progression-free survival (PFS).
Phase 1b: Assess Preliminary Efficacy in Terms of RECIST v1.1 for Immune Based Therapeutics | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine clinical benefit (complete response [CR] + partial response [PR] + stable disease [SD]).

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - UCLA, Los Angeles, California
  - Stanford, Stanford, California
  - University of Colorado, Denver, Colorado
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Washington University, Seattle, Washington